CLINICAL TRIAL: NCT05952882
Title: Effectiveness of the Combination Liraglutide and Metformin on Weight Loss, Metabolic - Endocrine Parameters and Pregnancy Rate in Women With Polycystic Ovarian Syndrome, Obesity and Infertility
Brief Title: Liraglutide and Metformin Combination on Weight Loss, Metabolic - Endocrine Parameters and Pregnancy Rate in Women With PCOS, Obesity and Infertility
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08/23/DD-BVMD
Record Dates: First submitted 2023-07-10; First posted 2023-07-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Polycystic Ovary Syndrome; Obesity; Infertility, Female
Keywords: Polycystic Ovary Syndrome; GLP-1 agonist; Liraglutide; obesity; weight loss; insulin resistance; androgens; pregnancy rates; In Vitro Fertilization
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Infertility, Female; Weight Loss; Insulin Resistance | interventions — Liraglutide; Metformin; lime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LIME 3mg/1500mg (Experimental): Metformin XR (extended-release) was initiated with a dose of 750 mg once per day for 2 week and increased to 1500 mg once per day for up to 12 weeks. Start injection liraglutide 0.6 mg subcutaneously (SC) 1week daily (QD), then titrated in increments of 0.6 mg once daily every 1 to 3 weeks to a final dose of 3.0 mg liraglutide SC daily for up to 12 weeks.
  Interventions: Drug: Liraglutide + Metformin
- MET 1500mg (Active Comparator): Metformin XR (extended-release) was initiated with a dose of 750 mg once per day for 2 week and increased to 1500 mg once per day for up to 12 weeks
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Liraglutide + Metformin — Metformin XR (extended-release) was initiated at 750 mg once daily and increased to 1500 mg once daily after 2 week. Concomitantly, Liraglutide was initiated at a subcutaneous dose of 0.6 mg once daily for 1 week, then titrated in increments of 0.6 mg once daily every 1 to 3 weeks to a maintenance dose of 3.0 mg once daily for up to 12 weeks
  Other Names: LIME
  Arms: LIME 3mg/1500mg
Drug: Metformin — Metformin XR (extended-release) was initiated at 750 mg once daily and increased to 1500 mg once daily after 2 week
  Other Names: MET
  Arms: MET 1500mg

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in women of reproductive age and one of the leading causes of infertility. PCOS and obesity affect up to 12.5% - 48.3% Asian women, increase incidence of impaired glucose tolerance, type 2 diabetes and aggravate insulin resistance, cause ovulatory dysfunction and menstrual disorders, and negatively impact outcomes of Assited Reproductive Technology (ART), with higher miscarriage rate when receiving ART. Weight loss decrease insulin resistance and hyperandrogenism, improve ovulation rate and menstrual cycle, significantly higher conception and live birth rates. Weight loss prior to IVF procedures has been associated with significantly improved pregnancy rates (PR) and live birth rates. Furthermore, a decreased number of IVF cycles required to achieve a pregnancy has also been reported after weight loss interventions. Based on the principles of fetal programming, improving a lifestyle before conception might lead to improved longterm health of the offspring. Studies on the effect of anti-obesity medication combined with lifestyle changes on body weight and composition and metabolic - endocrine parameters and pregnancy rate in obese women diagnosed with PCOS are lacking. There is a growing need to develop pharmacologic interventions to improve metabolic function in women with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
The drug, liraglutide 3.0 mg was approved for chronic weight management in management in obese adults with an initial BMI of 30 kg/m2 or greater or in overweight adults BMI of 27 kg/m2 or greater with at least one weight-related co-morbid condition as an adjunct to a reduced-calorie diet and increased physical activity. Liraglutide is an acylated human glucagon-like peptide -1 (GLP-1) analog that binds to and activates the GLP-1 receptor. It lowers body weight through decreased caloric intake while stimulating insulin secretion and reducing glucagon via a glucose-dependent mechanism. For obesity management, patients may lose weight with GLP-1 receptor agonists due to other unique actions. Glucagon-like peptide-1 receptor agonists (GLP-1RAs) can slow gastric emptying and increase satiety. While predictors of weight loss success for the general population are available (protein intake, weight loss medications), predictors of weight loss success may differ between normal and hyperandrogenic women. Glucagon-like peptide 1 agonists are linked with dose dependent weight lowering potential in different obesity related populations. The weight loss effects of GLP-1RAs previously demonstrated in diabetic and obese non-diabetic patients, offer a unique opportunity to expand the medical options available to patients with PCOS. Metformin was recommended for women with PCOS and obesity (BMI ≥ 25 kg/m2) or at metabolic risks and shown beneficial effects on menstrual disorders, anovulation, hyperandrogenism, and cardiovascular abnormalities.

The aim of this study was to evaluate the impact of liraglutide in combination with metformin compared to metformin alone on weight reduction, the multifaceted metabolic - endocrine disturbances, and oocyte and embryo quality, IVF PRs and cumulative PRs (IVF and spontaneous pregnancies) in infertile obese women with PCOS who had been previously poor responders to weight reduction with lifestyle modification.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* 18-65 years of age
* Diagnosis of polycystic ovary syndrome according to the revised Rotterdam criteria (2003)
* BMI ≥ 27 kg/m2
* Infertility
* Agree to participate in the study

Exclusion Criteria:

* Type 1 or type 2 diabetes.
* History of acute or chronic pancreatitis.
* Family or individual history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* Known hypersensitivity or contraindication to the use of GLP-1 receptor agonists.
* Used of hormonal drugs, drugs causing clinically significant weight changes and drugs affecting glucose tolerance for at least 8 weeks.
* Used a anti-androgen drugs for at least 4 weeks.
* History of malignancy requiring chemotherapy.
* History of taking antidiabetic drugs other than gestational diabetes or weight-loss drugs discontinued for at least 4 weeks.
* History of gastrectomy or device-based intervention to manage obesity
* Eating disorders (anorexia or bulimia) or digestive disorders.
* Substance abuse (Tobacco or alcohol)
* History of major depression or other serious mental disorder.
* Inability or refusal to adhere treatment regimens.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute Body Weight (BW) | 12 weeks of treatment
  Treatment impact on change in body weight after 12 weeks of treatment.
Change in Percent Body Weight | 12 weeks of treatment
  Treatment effect on reducing body weight expressed as percent body weight loss from baseline

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 12 weeks of treatment
  Treatment effect in reducing body mass
Abdominal Adiposity (Waist Circumference [WC]) | 12 weeks of treatment
  Treatment effect on loss of waist circumference (abdominal adiposity) with drug treatment
Waist-to-Hip Ratio (WHR) | 12 weeks of treatment
  Change in central adiposity with treatment as measured by waist-to-hip ratio. A reduction in ratio indicates a decrease in truncal fat.
Waist-to Height Ratio [WHtR] | 12 weeks of treatment
  Treatment effect on loss of central adiposity as determined by Waist-to Height Ratio. The lower the ratio indicates less abdominal adiposity.
Total Fat Mass Evaluated by BIA | 12 weeks of treatment
  Treatment effect on reduction of fat mass (kg)
Total Body Fat (%) by BIA (Bioelectrical Impedance Analysis) machine | 12 weeks of treatment
  Treatment effect on reduction of percent body fat by BIA
Visceral Fat Level (VFL) | 12 weeks of treatment
  Treatment effect on reduction of visceral fat level by BIA
Total lean body mass | 12 weeks of treatment
  Treatment impact on total lean body mass
Glucose OGTT 0 min | 12 weeks of treatment
  Treatment effect on fasting glucose prior to an oral glucose tolerance test (OGTT)
Glucose OGTT 120 min | 12 weeks of treatment
  Treatment effect on glucose measured at 120 minutes of an oral glucose tolerance test (OGTT)
Insulin OGTT 0 min | 12 weeks of treatment
  Treatment effect on fasting insulin prior to an oral glucose tolerance test (OGTT)
Insulin OGTT 120 min | 12 weeks of treatment
  Treatment effect on insulin measured at 120 minutes of an oral glucose tolerance test (OGTT)
Fasting Insulin Sensitivity (HOMA-IR) | 12 weeks of treatment
  Treatment effect on the HOMA-IR which is an insulin resistance measured derived from fasting blood glucose and insulin . The higher the number the more insulin resistant.
Matsuda Insulin Sensitivity Index Derived From the OGTT (SI OGTT) | 12 weeks of treatment
  The SI OGTT is a measure of peripheral insulin sensitivity derived from the insulin and glucoses measured during an OGTT. A increase in SI OGTTindicates greater insulin sensitivity
Total Cholesterol Levels | 12 weeks of treatment
  Treatment impact on improving total cholesterol levels
High Density Lipoprotein Cholesterol (HDL-C) | 12 weeks of treatment
  Impact of treatment on HDL levels after 12 weeks of treatment
Triglyceride Levels (TRG) | 12 weeks of treatment
  Drug effect of TRG levels after treatment
Low Density Lipoprotein Cholesterol (LDL-C) | 12 weeks of treatment
  Treatment impact on improving LDL-C after treatment
Systolic Blood Pressure | 12 weeks of treatment
  Treatment impact on systolic blood pressure
Diastolic Blood Pressure | 12 weeks of treatment
  Treatment impact on reducing diastolic blood pressure
Menstrual Cycle Frequency | 12 weeks of treatment
  Drug treatment impact on normalization of cycle frequency (cycle every 28-30 days). All cycle data is expressed as number of menses annualized to one year.
Free Androgen Index (FAI) | 12 weeks of treatment
  Drug treatment effect on free androgen levels as calculated as FAI= total testosterone (T) concentrations divided by sex hormone binding globulin (SHBG) levels. A higher score indicates a worse outcome (more androgenic).
Total Testosterone Concentrations (T) | 12 weeks of treatment
  Drug treatment effect on total testosterone concentrations
Sex Hormone Binding Globulin (SHBG) | 12 weeks of treatment
  Drug treatment effect on SHBG
Adrenal Dehydroepiandrosterone Sulfate (DHEAS) | 12 weeks of treatment
  Treatment efficacy in reducing adrenal hyperandrogenism
17(OH)-progesterone | 12 weeks of treatment
  Treatment efficacy in reducing adrenal hyperandrogenism
Androstenedione | 12 weeks of treatment
  Drug treatment effect on androstenedione
Progesterone | 12 weeks of treatment
  Drug treatment effect on progesterone
Luteinizing Hormone (LH) | 12 weeks of treatment
  Drug treatment effect on LH
Follicle Stimulating Hormone (FSH) | 12 weeks of treatment
  Drug treatment effect on FSH
Ovary Volume | 12 weeks of treatment
  Treatment efficacy in reducing ovary volume
Spontaneous Pregnancy Rate | 12 months after treatment
  Treatment effect on spontaneous pregnancy rate
Assisted Reproductive Therapy Pregnancy Rate | 12 months after treatment
  Treatment effect on Assisted Reproductive Therapy Pregnancy Rate
Cumulative Pregnancy Rate | 12 months after treatment
  Treatment effect on Cumulative Pregnancy Rate
Total dosage gonadotropin (GNT) | 12 weeks of treatment
  Drug treatment impact on total dosage GNT
No. of retrieved oocytes/patient | 12 weeks of treatment
  Drug treatment impact on No. of retrieved oocytes/patient
No. of mature (MII) oocytes/patient | 12 weeks of treatment
  Drug treatment impact on No. of mature (MII) oocytes/patient
Fertilization rate | 12 weeks of treatment
  Drug treatment impact on fertilization rate
Oocyte degeneration rate | 12 weeks of treatment
  Drug treatment impact on oocyte degeneration rate
Immaturity rate | 12 weeks of treatment
  Drug treatment impact on immaturity rate
No. of embryos on day 5/patient | 12 weeks of treatment
  Drug treatment impact on No. of embryos on day 5/patient
No. of blastocysts/patient | 12 weeks of treatment
  Drug treatment impact on No. of blastocysts/patient
Blastulation rate | 12 weeks of treatment
  Drug treatment impact on blastulation rate
No. of transferred embryos | 12 weeks of treatment
  Drug treatment impact on No. of transferred embryos
Pregnancy rate per cycle | 12 weeks of treatment
  Drug treatment impact on pregnancy rate per cycle
Pregnancy rate per Embryo Transfer (ET) | 12 weeks of treatment
  Drug treatment impact on pregnancy rate per ET
Implantation rate | 12 weeks of treatment
  Drug treatment impact on implantation rate
No. of cancelled fresh Embryo Transfer (ET) because of hyperstimulation risk | 12 weeks of treatment
  Drug treatment impact on No. of cancelled fresh Embryo Transfer (ET because of hyperstimulation risk
Cryopreservation | 12 weeks of treatment
  Drug treatment impact on cryopreservation
No. of cryopreserved embryos/patient | 12 weeks of treatment
  Drug treatment impact on No. of cryopreserved embryos/patient
Ectopic Pregnancy Rate | 12 weeks of treatment
  Drug treatment impact on Ectopic Pregnancy Rate
Stillbirth Rate | 24 months after treatment
  Drug treatment impact on Stillbirth Rate
Abortion Rate | 24 months after treatment
  Drug treatment impact on Abortion Rate
Gestational Diabetes Mellitus Rate | 24 months after treatment
  Drug treatment impact on Gestational Diabetes Mellitus Rate
Gestational hypertensive disorder (GHD) Rate | 24 months after treatment
  Drug treatment impact on Gestational hypertensive disorder (GHD) Rate
Live Birth Rate | 24 months after treatment
  Drug treatment impact on Live Birth Rate
Gestational age at birth | 24 months after treatment
  Drug treatment impact on gestational age at birth
Type of Delivery Method | 24 months after treatment
  Drug treatment impact on Type of Delivery Method

REFERENCES:
- [Result] Rosenfield RL, Ehrmann DA. The Pathogenesis of Polycystic Ovary Syndrome (PCOS): The Hypothesis of PCOS as Functional Ovarian Hyperandrogenism Revisited. Endocr Rev. 2016 Oct;37(5):467-520. doi: 10.1210/er.2015-1104. Epub 2016 Jul 26. PMID 27459230
- [Result] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Result] Lim SS, Davies MJ, Norman RJ, Moran LJ. Overweight, obesity and central obesity in women with polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod Update. 2012 Nov-Dec;18(6):618-37. doi: 10.1093/humupd/dms030. Epub 2012 Jul 4. PMID 22767467
- [Result] Zeng X, Xie YJ, Liu YT, Long SL, Mo ZC. Polycystic ovarian syndrome: Correlation between hyperandrogenism, insulin resistance and obesity. Clin Chim Acta. 2020 Mar;502:214-221. doi: 10.1016/j.cca.2019.11.003. Epub 2019 Nov 13. PMID 31733195
- [Result] Norman RJ, Masters L, Milner CR, Wang JX, Davies MJ. Relative risk of conversion from normoglycaemia to impaired glucose tolerance or non-insulin dependent diabetes mellitus in polycystic ovarian syndrome. Hum Reprod. 2001 Sep;16(9):1995-8. doi: 10.1093/humrep/16.9.1995. PMID 11527911
- [Result] Dunaif A, Segal KR, Futterweit W, Dobrjansky A. Profound peripheral insulin resistance, independent of obesity, in polycystic ovary syndrome. Diabetes. 1989 Sep;38(9):1165-74. doi: 10.2337/diab.38.9.1165. PMID 2670645
- [Result] Practice Committee of the American Society for Reproductive Medicine. Electronic address: asrm@asrm.org; Practice Committee of the American Society for Reproductive Medicine. Obesity and reproduction: a committee opinion. Fertil Steril. 2021 Nov;116(5):1266-1285. doi: 10.1016/j.fertnstert.2021.08.018. Epub 2021 Sep 25. PMID 34583840
- [Result] Zhang J, Liu H, Mao X, Chen Q, Fan Y, Xiao Y, Wang Y, Kuang Y. Effect of body mass index on pregnancy outcomes in a freeze-all policy: an analysis of 22,043 first autologous frozen-thawed embryo transfer cycles in China. BMC Med. 2019 Jun 26;17(1):114. doi: 10.1186/s12916-019-1354-1. PMID 31238940
- [Result] Metwally M, Ong KJ, Ledger WL, Li TC. Does high body mass index increase the risk of miscarriage after spontaneous and assisted conception? A meta-analysis of the evidence. Fertil Steril. 2008 Sep;90(3):714-26. doi: 10.1016/j.fertnstert.2007.07.1290. Epub 2008 Feb 6. PMID 18068166
- [Result] Panidis D, Farmakiotis D, Rousso D, Kourtis A, Katsikis I, Krassas G. Obesity, weight loss, and the polycystic ovary syndrome: effect of treatment with diet and orlistat for 24 weeks on insulin resistance and androgen levels. Fertil Steril. 2008 Apr;89(4):899-906. doi: 10.1016/j.fertnstert.2007.04.043. Epub 2007 Nov 5. PMID 17980364
- [Result] Legro RS, Dodson WC, Kris-Etherton PM, Kunselman AR, Stetter CM, Williams NI, Gnatuk CL, Estes SJ, Fleming J, Allison KC, Sarwer DB, Coutifaris C, Dokras A. Randomized Controlled Trial of Preconception Interventions in Infertile Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2015 Nov;100(11):4048-58. doi: 10.1210/jc.2015-2778. Epub 2015 Sep 24. PMID 26401593
- [Result] Best D, Avenell A, Bhattacharya S. How effective are weight-loss interventions for improving fertility in women and men who are overweight or obese? A systematic review and meta-analysis of the evidence. Hum Reprod Update. 2017 Nov 1;23(6):681-705. doi: 10.1093/humupd/dmx027. PMID 28961722
- [Result] Kort JD, Winget C, Kim SH, Lathi RB. A retrospective cohort study to evaluate the impact of meaningful weight loss on fertility outcomes in an overweight population with infertility. Fertil Steril. 2014 May;101(5):1400-3. doi: 10.1016/j.fertnstert.2014.01.036. Epub 2014 Feb 26. PMID 24581574
- [Result] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Fertil Steril. 2018 Aug;110(3):364-379. doi: 10.1016/j.fertnstert.2018.05.004. Epub 2018 Jul 19. PMID 30033227
- [Result] Legro RS, Arslanian SA, Ehrmann DA, Hoeger KM, Murad MH, Pasquali R, Welt CK; Endocrine Society. Diagnosis and treatment of polycystic ovary syndrome: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2013 Dec;98(12):4565-92. doi: 10.1210/jc.2013-2350. Epub 2013 Oct 22. PMID 24151290
- [Result] Palomba S, Falbo A, Zullo F, Orio F Jr. Evidence-based and potential benefits of metformin in the polycystic ovary syndrome: a comprehensive review. Endocr Rev. 2009 Feb;30(1):1-50. doi: 10.1210/er.2008-0030. Epub 2008 Dec 4. PMID 19056992
- [Result] Dunaif A. Drug insight: insulin-sensitizing drugs in the treatment of polycystic ovary syndrome--a reappraisal. Nat Clin Pract Endocrinol Metab. 2008 May;4(5):272-83. doi: 10.1038/ncpendmet0787. Epub 2008 Mar 25. PMID 18364705
- [Result] Diamanti-Kandarakis E, Christakou CD, Kandaraki E, Economou FN. Metformin: an old medication of new fashion: evolving new molecular mechanisms and clinical implications in polycystic ovary syndrome. Eur J Endocrinol. 2010 Feb;162(2):193-212. doi: 10.1530/EJE-09-0733. Epub 2009 Oct 19. PMID 19841045
- [Result] Abdalla MA, Deshmukh H, Atkin S, Sathyapalan T. The potential role of incretin-based therapies for polycystic ovary syndrome: a narrative review of the current evidence. Ther Adv Endocrinol Metab. 2021 Jan 27;12:2042018821989238. doi: 10.1177/2042018821989238. eCollection 2021. PMID 33552465
- [Result] Knudsen LB, Lau J. The Discovery and Development of Liraglutide and Semaglutide. Front Endocrinol (Lausanne). 2019 Apr 12;10:155. doi: 10.3389/fendo.2019.00155. eCollection 2019. PMID 31031702
- [Result] Cena H, Chiovato L, Nappi RE. Obesity, Polycystic Ovary Syndrome, and Infertility: A New Avenue for GLP-1 Receptor Agonists. J Clin Endocrinol Metab. 2020 Aug 1;105(8):e2695-709. doi: 10.1210/clinem/dgaa285. PMID 32442310
- [Result] Han Y, Li Y, He B. GLP-1 receptor agonists versus metformin in PCOS: a systematic review and meta-analysis. Reprod Biomed Online. 2019 Aug;39(2):332-342. doi: 10.1016/j.rbmo.2019.04.017. Epub 2019 Apr 25. PMID 31229399
- [Result] Frossing S, Nylander M, Chabanova E, Frystyk J, Holst JJ, Kistorp C, Skouby SO, Faber J. Effect of liraglutide on ectopic fat in polycystic ovary syndrome: A randomized clinical trial. Diabetes Obes Metab. 2018 Jan;20(1):215-218. doi: 10.1111/dom.13053. Epub 2017 Aug 11. PMID 28681988
- [Result] Jensterle Sever M, Kocjan T, Pfeifer M, Kravos NA, Janez A. Short-term combined treatment with liraglutide and metformin leads to significant weight loss in obese women with polycystic ovary syndrome and previous poor response to metformin. Eur J Endocrinol. 2014 Feb 7;170(3):451-9. doi: 10.1530/EJE-13-0797. Print 2014 Mar. PMID 24362411
- [Result] Nylander M, Frossing S, Clausen HV, Kistorp C, Faber J, Skouby SO. Effects of liraglutide on ovarian dysfunction in polycystic ovary syndrome: a randomized clinical trial. Reprod Biomed Online. 2017 Jul;35(1):121-127. doi: 10.1016/j.rbmo.2017.03.023. Epub 2017 Apr 24. PMID 28479118
- [Result] Salamun V, Jensterle M, Janez A, Vrtacnik Bokal E. Liraglutide increases IVF pregnancy rates in obese PCOS women with poor response to first-line reproductive treatments: a pilot randomized study. Eur J Endocrinol. 2018 Jul;179(1):1-11. doi: 10.1530/EJE-18-0175. Epub 2018 Apr 27. PMID 29703793
- [Result] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Fertil Steril. 2017 Sep;108(3):393-406. doi: 10.1016/j.fertnstert.2017.06.005. Epub 2017 Jul 29. PMID 28760517